CLINICAL TRIAL: NCT05639400
Title: Thoraflex Hybrid and Relay Extension Post-Approval Study
Acronym: EXTEND
Status: Active, not recruiting | Type: Observational
Sponsor: Vascutek Ltd. (Industry)
Collaborators: Bolton Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: EXTEND-001
Record Dates: First submitted 2022-11-24; First posted 2022-12-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thoracic Diseases; Aortic Aneurysm; Aortic Dissection; Thoracic Aortic Aneurysm; Thoracic Aortic Dissection
Keywords: TEVAR; Frozen Elephant Trunk (FET)
MeSH Terms: conditions — Thoracic Diseases; Aortic Aneurysm; Aortic Dissection; Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Thoraflex Hybrid — Thoraflex Hybrid is designed for the open surgical repair of aneurysms and/or dissections in the aortic arch and descending aorta with or without involvement of the ascending aorta. There are two types of Thoraflex Hybrid implants, namely the Plexus 4 and the Ante-Flo versions. Each patient receives one Thoraflex Hybrid device (either the Plexus 4 or Ante-Flo).
Device: RelayPro NBS — The RelayPro NBS Thoracic Stent-Graft System is an endovascular device intended for treatment of thoracic aortic pathologies such as aneurysms, pseudoaneurysms, dissections, penetrating ulcers and intramural hematoma.

SUMMARY:
The goal of this observational study is to evaluate the Thoraflex Hybrid device alone and in combination with the RelayPro NBS stent-graft in the treatment of aortic disease affecting the aortic arch and descending aorta with or without involvement of the ascending aorta.

Patients who undergo treatment with the Thoraflex Hybrid device with or without extension with a RelayPro NBS stent-graft will be eligible for enrolment and study activities and follow-up regime will follow standard care at each participating site.

Participant involvement in the study will last for a total of 10 years from the point at which the Thoraflex Hybrid device is placed.

ELIGIBILITY:
Inclusion Criteria:

Patient is aged 18 years or older on date of consent. Patient is willing and able to comply with all study procedures and visits. Patient or their next of kin (NOK)/legally designated representative (LDR) has given written informed consent to participate in the study.

Patient will undergo treatment with a Thoraflex Hybrid device. If a patient requires an extension procedure due to the extent of aortic disease, a RelayPro NBS Stent-graft should be placed inside the distal end of the previously placed Thoraflex Hybrid device via a retrograde approach. This may be part of the same or a two-stage procedure.

Exclusion Criteria:

* Patient has any medical, social, or psychological problems that in the opinion of the investigator preclude them from receiving this treatment and the procedures and evaluations pre and post procedure.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who undergo treatment with the Thoraflex Hybrid device with or without extension with a RelayPro NBS stent-graft.
Sampling Method: Probability Sample
Enrollment: 352 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2036-03 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint is a composite of the following: | The primary safety endpoint will be measured at one-year after the index procedure and again at least 8 months after the (first) extension procedure.
  * Permanent disabling stroke (mRS >2 and an increase in at least one mRS category from the individual's pre-stroke baseline, occurring within 30 days of either index procedure or extension and present at 1-year follow-up)* Note: If a subject dies prior to 1-year follow-up, their last recorded mRS will be considered their final score
  * Grade 3 spinal cord ischemia (SVS reporting standards) occurring within 30 days of either index procedure or extension
  * All-cause mortality (within 1 year of either procedure)
  (*Per VARC-3, disability assessment using the mRS should be performed between 30 and 90 days after a neurological event with 90 days being optimal. An increased mRS score by itself and in the absence of a neurological event does not constitute stroke.)
Primary Effectiveness Endpoint: Treatment Success | The primary effectiveness endpoint will be measured at one-year after the index procedure and again at least 8 months after the (first) extension procedure.
  Defined as device technical success (of either procedure) with absence of the following at 1-year:
  * Lesion-related mortality (defined as all deaths occurring within 30 days of, or, prior to discharge, from either the index procedure or the extension procedure or any revision procedures to treat the original lesion(s) and any other deaths adjudicated by Clinical Events Committee as related or probably related to the lesion(s))
  * Aortic rupture in the treated segment
  * Lesion expansion (≥5mm increase from measurement at discharge/within 30 days)
  * Secondary intervention to address the following:
    * Stent graft-induced aortic wall injury (SAWI)
    * Fistula
    * Type I or III endoleak (see definitions)
    * Migration
    * Loss of Patency
    * Thromboembolic events
    * Failure of integrity

SECONDARY OUTCOMES:
Secondary Safety Endpoints, Absence of the following | The secondary endpoints will be measured at each follow-up timepoint from discharge/30 days through to 10 years.
  * All-cause mortality, and
  * Lesion-related mortality (defined as all deaths occurring within 30 days of, or, prior to discharge, from either the index procedure or the extension procedure or any revision procedures to treat the original lesion(s) and any other deaths adjudicated by Clinical Events Committee as related or probably related to the lesion(s))
  * All/any paraplegia/paraparesis defined as SCI (SVS grades 1 to 3)
  * Any stroke (excluding TIA)
  * Incidence of Myocardial Infarction
  * Incidence of Respiratory Failure
  * Incidence of Renal Failure
  * Incidence of Bowel Ischemia
Secondary effectiveness endpoints will be reported | The secondary endpoints will be measured at each follow-up timepoint from discharge/30 days through to 10 years.
  * Any aortic rupture (treated and untreated segments)
  * Aortic remodeling in the treated segment(s)
  * New dissections
  * Proximal and distal extension of dissections
  * Any false lumen perfusion (specifying location and if intentional or not)
  * Fistula formation
  * All endoleaks
  * Device migration (measure both >5mm from position at discharge/within 30 days, and >10 mm from position at discharge/within 30 days, and requiring secondary intervention)
  * Device integrity issues (e.g., stent fracture)
  * All thromboembolic events
  * Pseudoaneurysms (device-related)
  * Secondary Interventions
  * Graft patency (loss of patency will be defined as an opening of <50% due to, for example, occlusion, stenosis, kinking)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Czerny, Principal Investigator — University of Freiburg; Joseph E Bavaria, Principal Investigator — Jefferson Health and Sidney Kimmel Medical College
Locations (27):
- United States (18):
  - University of Alabama in Birmingham Medical Center, Birmingham, Alabama
  - Cedars-Sinai Medical Centre, Los Angeles, California
  - Keck Medical Centre of USC, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Medstar Washington Hospital Centre, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Ascension St. Vincent Heart Center, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - Weill Cornell medicine, New York, New York
  - Duke University Medical Centre, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UT Dell Medical / Ascension Texas Cardiovascular, Austin, Texas
  - Baylor College of Medicine - St. Luke's, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Paracelsus Medical University, Salzburg, Austria
- France (2):
  - CHU Nantes, Saint-Herblain
  - CHU de Toulouse - Hôpital de Rangueil, Toulouse
- University of Freiburg, Freiburg im Breisgau, Germany
- Policlinico Di S.Orsola, Universita' Di Bologna, Bologna, Italy
- Hospital Clinic of Barcelona, Barcelona, Spain
- United Kingdom (3):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Oxford University Hospitals NHS FT, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Undecided